CLINICAL TRIAL: NCT04021914
Title: Demonstrating Feasibility of Color Vision Deficient Provider Use of EnChroma Products in the Emergency Department
Brief Title: Feasibility of EnChroma Use in the Emergency Department Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment and study activities were terminated due to difficulties with recruitment of participants.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jeffrey Siegelman, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00111894
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Color Vision Defects
Keywords: CVD; color vision deficiency; healthcare providers; emergency department; Enchroma glasses
MeSH Terms: conditions — Color Vision Defects; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EnChroma glasses (Experimental): EnChroma products improve brightness and color purity of primary colors for CVD people. Each participant with CVD will be provided EnChroma products to use indoors over the course of two weeks in the emergency department, educational settings, and in their personal life.
  Interventions: Device: EnChroma glasses

INTERVENTIONS:
Device: EnChroma glasses — Each participant will be provided EnChroma products to use indoors over the course of two weeks in the emergency department, educational settings, and in their personal life. They will be encouraged to wear the glasses for at least 10 hours over 1-2 weeks prior to wearing them in a clinical setting to adjust to their use, and for 10 minutes before beginning patient care as per manufacturer instructions. They will be encouraged to take specific note of clinical scenarios that require the use of color vision (e.g., - rashes, tympanic membrane erythema, stool guaiac testing, etc.).

SUMMARY:
This study addresses whether the use of EnChroma products are feasible for use in the emergency department by color vision deficient providers.

DETAILED DESCRIPTION:
This study addresses whether it is feasible for color vision deficient (CVD) physicians and other healthcare providers to wear EnChroma products in the clinical setting. It is known that color vision is important to the practice of medicine. Identifying red skin or red ear drums, noticing whether lips have turned blue or a patient is pale, and identifying colors under a microscope all are aided by or dependent upon color vision. While color vision deficiency does not preclude a person from becoming and succeeding as a physician, it may be appropriate and desired to utilize devices to improve color vision during patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Red-Green color deficiency

Exclusion Criteria:

* Achromatopsia
* Cataracts
* Glaucoma
* Legal blindness
* Macular degeneration
* Retinitis Pigmentosa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Siegelman, MD, Principal Investigator — Emory Univer
Locations (1):
- Emory Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between August 2019 and March 2023.
Period: Overall Study
Arm/Group | EnChroma Glasses
Started | 6
Completed | 5
Not Completed | 1
Not completed — Did not meet inclusion criteria on confirmatory testing | 1

BASELINE CHARACTERISTICS:
Population: Participants who signed the consent and started study activities.
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Color Vision Perception Based on Patients' Description
Description: Subjective influence of EnChroma glasses will be assessed by asking to describe a difference that the glasses made in color vision. The overall quality of color perception will be assessed with a scale from 1 to 10. Higher score correlates highest quality (better outcome).
Time Frame: 2 weeks post-intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
score on a scale | 6.5 (1.7)

2. Primary Outcome: Overall Quality of Color Vision Perception in Normal Daylight Based on Patients' Description
Description: Subjective influence of EnChroma glasses will be assessed by asking to describe a difference that the glasses made in color vision perception in normal daylight based on patients' description. The overall quality of color perception will be assessed with a scale from 1 to 10. Higher score correlates highest quality (better outcome).
Time Frame: 2 weeks post-intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
score on a scale | 7 (1.8)

3. Primary Outcome: Overall Quality of Color Vision Perception in Dim Light Based on Patients' Description
Description: Subjective influence of EnChroma glasses will be assessed by asking to describe a difference that the glasses made in color vision perception in dim light based on patients' description. The overall quality of color perception will be assessed with a scale from 1 to 10. Higher score correlates highest quality (better outcome).
Time Frame: 2 weeks post-intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
score on a scale | 5.5 (2.5)

4. Primary Outcome: Number of Participants Reporting More Positive Than Negative Comments About the Use of the EnChroma Glasses
Description: Comfort of EnChroma glasses will be assessed by a multiple choice question, where a respondent can choose from listed negative or positive responses (e.g., did or didn't like, comfortable or uncomfortable, ). Number of participants reporting more positive than negative comments about the use of the EnChroma glasses will be reported.
Time Frame: 2 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Number of Participants That Reported an Impact of Using the Glasses on Patient Care
Description: Number of participants that reported an impact of the glasses on patient care, especially in situations that require the use of color vision (e.g., - rashes, tympanic membrane erythema, stool guaiac testing, etc.), will be assessed by asking a question. Participants that report impact is associated with better outcome.
Time Frame: 2 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | EnChroma Glasses
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Time Frame: All adverse events were collected and documented during the duration of study participation= two (2) weeks
Arm/Group | EnChroma Glasses
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04021914/Prot_SAP_000.pdf